CLINICAL TRIAL: NCT02802514
Title: An Exploratory Randomized, 2-Part, Single-blind, 2-Period Crossover Study Comparing the Effect of Albiglutide With Exenatide on Regional Brain Activity Related to Nausea in Healthy Volunteers
Brief Title: A Study Comparing the Effect of Albiglutide With Exenatide on Regional Brain Activity Related to Nausea in Healthy Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: The General Hospital Corporation d/b/a Massachusetts General Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 201840
Record Dates: First submitted 2016-06-02; First posted 2016-06-16 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus
Keywords: Gastrointestinal; Glucagon like peptide; Nausea; Magnetic resonance imaging
MeSH Terms: conditions — Diabetes Mellitus; Nausea | interventions — rGLP-1 protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- With Off therapy MRI in S1:Albiglutide-S1 & Exenatide-S2 (Experimental): In session 1, eligible subject will undergo off-therapy MRI scan Subject will receive single dose each of 50 mg albiglutide on Day 5 and exenatide placebo on Day 8 followed by a post-dose MRI. In session 2, subject will receive single dose each of albiglutide placebo on Day 1 (Week 9) and 10 microgram exenatide on Day 4 followed by a post-dose MRI scan. There will be 6-9 week washout period between Session 1 and Session 2
  Interventions: Drug: Albiglutide 50mg; Drug: Albiglutide matching placebo; Drug: Exenatide 10microgram; Drug: Exenatide placebo (saline)
- Without Off therapy MRI in S1:Albiglutide-S1 & Exenatide-S2 (Experimental): In session 1, eligible subject will receive single dose each of 50 mg albiglutide on Day 1 and exenatide placebo on Day 4 followed by a post-dose MRI scan. In session 2, Day 1 (Week 9) subject will undergo off-therapy MRI scan. Subject will receive single dose each of albiglutide placebo on Day 5 and 10 microgram of exenatide on Day 8 followed by a post-dose MRI scan. There will be 6-9 week washout period between Session 1 and Session 2
  Interventions: Drug: Albiglutide 50mg; Drug: Albiglutide matching placebo; Drug: Exenatide 10microgram; Drug: Exenatide placebo (saline)
- With Off therapy MRI in S1:Exenatide-S1 & Albiglutide-S2 (Experimental): In session 1, Day 1 subject will undergo off-therapy MRI scan Subject will receive single dose each of albiglutide placebo on Day 5 and 10 microgram of exenatide on Day 8 followed by a post-dose MRI scan In session 2, eligible subject will receive single dose each of 50 mg albiglutide on Day 1 (Week 9) and exenatide placebo Day 4 followed by a post-dose MRI scan. There will be 6-9 week washout period between Session 1 and Session 2
  Interventions: Drug: Albiglutide 50mg; Drug: Albiglutide matching placebo; Drug: Exenatide 10microgram; Drug: Exenatide placebo (saline)
- Without Off therapy MRI in S1: Exenatide-S1 & Albiglutide-S2 (Experimental): In session 1, subject will receive single dose each of albiglutide placebo on Day 1 and 10 microgram exenatide on Day 4 followed by a post-dose MRI scan. In session 2, subject will undergo off-therapy MRI scan on Day 1 (Week 9). Subject will receive single dose each of 50 mg albiglutide on Day 5 and exenatide placebo on Day 8 followed by a post-dose MRI scan.. There will be 6-9 week washout period between Session 1 and Session 2
  Interventions: Drug: Albiglutide 50mg; Drug: Albiglutide matching placebo; Drug: Exenatide 10microgram; Drug: Exenatide placebo (saline)

INTERVENTIONS:
Drug: Albiglutide 50mg — It is provided as a single use fixed dose disposable pen injector (0.5 mL) system for SC delivery. A 50 mg pen contains 67 mg lyophilized albiglutide and 0.65 mL diluents. It will be injected subcutaneously (SC) in the upper arm.
Drug: Albiglutide matching placebo — It is provided as a single use fixed dose disposable pen injector (0.5 mL) system for SC delivery. It will be injected subcutaneously (SC) in the upper arm
Drug: Exenatide 10microgram — It is provided as a sterile solution containing 250 microgram/mL exenatide. One dose of 10 microgram is equivalent to 0.04 ml. It will be injected subcutaneously (SC) in the upper arm
Drug: Exenatide placebo (saline) — It is provided as a sterile saline. It will be injected subcutaneously (SC) in the upper arm

SUMMARY:
The drug effects will be studied after a single dose of 50 milligram (mg) albiglutide and a single dose of 10 microgram exenatide, to gain insight into the central mechanisms of nausea associated with Glucagon-like peptide-1 receptor (GLP-1R) agonists. This study will explore the potential differences at the expected time of maximum concentration (Cmax) between a long-acting (albiglutide) and short-acting (exenatide) GLP-1R agonist in brain activation of healthy volunteers assessed by magnetic resonance imaging (MRI). This is a phase IV, 2-part, 2-period crossover (session), single dose, randomized, single blind (blinded to both the subject and the imaging evaluators analysing the MRI data), placebo- and active-controlled study in adult healthy volunteers who are susceptible to motion sickness. Part A and Part B are the same in design, both consisting of a screening stage, a dosing/assessment stage, and a follow-up visit. Data from Part A will inform progression, methods, and analysis plan for Part B. Each sequence includes three scanning visits: albiglutide plus scan, exenatide plus scan and an off-therapy -natural history scan with a 6-9 week washout period between the dosing scans. A total of 24 to 28 subjects will be randomized in the study (Part A and Part B). The cross over design is divided into 2 sessions and schedule is as follow, on Day 1 (either Session 1 (S1) or Session 2 (S2) per, if randomized) subject will under go an off-therapy MRI scan, on Day 5 subject will receive a single dose of 50 mg albiglutide or albiglutide placebo, and Day 8 subject will receive a single dose of 10 microgram exenatide or saline placebo followed by a post-dose MRI scan. At each session subject will receive only one active drug (albiglutide or exenatide).

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Pure right-handed based on Edinburgh Handedness Inventory
* Motion Sickness Susceptibility Questionnaire (MSSQ) Screening score >60 and mock fMRI nausea rating >=2
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator (in consultation with the Medical Monitor, if necessary) decides and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or ability to interpret study results.
* Subject's body mass index (BMI) is >=19 (kilogram per square meter)kg/m^2 and =<30 kg/m^2
* Male OR
* Female: eligible to participate if she is not pregnant (as confirmed by a negative human chorionic gonadotrophin (hCG) test at screening and at other timepoints), not lactating, and at least one of the following conditions applies: a. Non-reproductive potential defined as pre-menopausal females who are having documented tubal ligation or Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or hysterectomy or documented Bilateral Oophorectomy OR Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause to confirm (refer to laboratory reference ranges for confirmatory levels)]. b. Reproductive potential and agrees to follow one of the options listed for avoiding pregnancy in females of reproductive potential (FRP) requirements from 30 days prior to the first dose of study medication and for the duration of study including the completion of the follow-up visit. The options are, Contraceptive subdermal implant or Intrauterine device or intrauterine system or Combined estrogen and progestogen oral contraceptive or Injectable progestogen or Contraceptive vaginal ring or Percutaneous contraceptive patches or Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject. The documentation on male sterility can come from the site personnel's: review of subject's medical records, medical examination and/or semen analysis, or medical history interview provided by her or her partner.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions.

Exclusion Criteria:

* Severe nausea (with or without vomiting) in the last three months or any event of unexplained nausea (with or without vomiting) as reported by the subject in the last 14 days before screening.
* History of vestibular or balance disorders as determined by the Investigator.
* History of smoking cigarettes or using tobacco products or any nicotine-containing products (including nicotine patches) within 3 months of screening.
* Use of eyeglasses during functional MRI (fMRI). Subjects requiring visual correction to participate in visual task that cannot be corrected with contact lenses.
* Alanine amino transferase (ALT) >1.5xupper limit of normal (ULN)
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 msec
* Systolic blood pressure is >=140 millimeter of Mercury (mm Hg) at Screening; repeat blood pressures should be taken if the subject's systolic blood pressure is >=140 mm Hg and if the results are consistently >=140 mm Hg, then the subject will be excluded and advised to consult a physician
* Diastolic blood pressure is >=90 mm Hg at Screening; repeat blood pressures should be taken if the subject's diastolic blood pressure is >=90 mm Hg and if the results are consistently >=90 mm Hg, then the subject should be excluded and advised to consult a physician
* Mean resting heart rate is >100 beats/minutes (mins) out of 3 consecutive measures taken 10 mins apart at Screening
* History of intestinal obstruction, ileus, gastrointestinal surgery or any other medical condition or procedure (e.g., gastrectomy, gastric bypass, lap-band) that may impair gastrointestinal motility
* History of significant cardiovascular or pulmonary dysfunction prior to screening
* History of acute or chronic pancreatitis
* History of severe gastrointestinal disease, including gastroparesis, inflammatory bowel disease, Crohn's disease, or irritable bowel syndrome
* History of any significant psychiatric illness (e.g., schizophrenia, bipolar affective disorder, bulimia or anorexia nervosa) that in the opinion of the Investigator would interfere with participation in the study.
* History and/or evidence of any other Central Nervous System (CNS) disorder that in the opinion of the Investigator would interfere with participation in the study (e.g., epilepsy, brain tumour, brain surgery).
* History of clinically significant CNS trauma (e.g. traumatic brain injury, cerebral contusion, spinal cord compression) or seizures.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Received within 7 days prior to screening or unable to refrain from taking for the duration of each part of study, medications that might; modify gastric myoelectical activity or gastrointestinal motility as prokinetic (e.g., erythromycin), anti-emetic agents (e.g., metoclopromide), narcotic analgesics (e.g., morphine), anticholinergic drugs (e.g., domperidone), anti-acid (e.g., pump inhibitors, H2 blockers) and laxative agents or
* stimulate or inhibit CNS (e.g., modafinil, dexamphetamine, methylphenidate, bromopheniramine, chlorpheniramine, clemastine, diphenhydramine, hyrdoxyzine)
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Is unwilling to abstain from alcohol for 24 hours before dosing and before each MRI scanning visit
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Subject has a history of significant weight loss (>5% reported change within 3 months prior to screening) or is currently attempting weight loss
* History of hypersensitivity to albiglutide, exenatide, or any product components
* Personal or family history of multiple endocrine neoplasia type 2, or medullary carcinoma of the thyroid
* Subject has any known condition(s) that may be contraindicated or interfere with the completion of MRI scanning such as implants (e.g., pacemaker, cochlear), a medical or electronic device (e.g., metallic joint prostheses, metal pins, screws, plates, stents or surgical staples), or claustrophobia.
* An abnormal (i.e., outside the normal reference range) thyroid function test assessed by thyroid stimulating hormone and Free T4 at screening.
* An abnormal amylase or lipase test at screening
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening or at screening
* A positive pre-study drug/alcohol screen
* A positive test for human immunodeficiency virus (HIV) antibody
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56-day period
* Subject has previously received any Glucagon-like peptide-1 receptor (GLP-1R) agonist at any time (e.g., albiglutide, exenatide, liraglutide, lixisenatide, dulaglutide)
* Subject has previously received dipeptidyl peptidase 4 (DPP-IV) inhibitor (sitagliptin, saxagliptin, linagliptin, alogliptin) within 30 days from screening
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 new investigational products within 12 months prior to the first dosing day

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This crossover study conducted in adult healthy volunteers who were susceptible to motion sickness to explore regional brain activity and connectivity associated with treatment using magnetic resonance imaging (MRI). Participants were randomized to receive single dose of 50milligram (mg) albiglutide and 10microgram (µg) exenatide along with placebo
Pre-assignment Details: A total of 10 participants were screened, of which 6 were screen-failures and 4 were randomized. Participants from United States site were part of the study. This was a 2-part study; however, study was terminated early due to portfolio strategic reason and only Part A was completed.
Groups:
- Session 1 Off-therapy MRI+Albiglutide Followed by Session 2: Participants underwent off-therapy MRI on Day 1 then received albiglutide 50 mg on Day 5 followed by exenatide matching placebo on Day 8 during Session 1. Post-dose MRI was conducted following exenatide placebo on Day 8 in session 1. There was a wash-out period of 6-9 weeks between the two sessions. In Session 2 participants received albiglutide matching placebo on Day 1 followed by 10 µg of exenatide on Day 4. Post-dose MRI was conducted following exenatide dose on Day 4 in session 2. Placebo was used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind. Hence, post-exenatide placebo MRI served as the post-albiglutide MRI in this study, to preserve the study blinding and to allow albiglutide sufficient time to reach Tmax.
- Session 1 Off-therapy MRI+Exenatide Followed by Session 2: Participants underwent off-therapy MRI on Day 1 then received albiglutide matching placebo on Day 5 followed by 10 µg of exenatide on Day 8 during Session 1. Post-dose MRI was conducted following exenatide dose on Day 8 in session 1. There was a wash-out period of 6-9 weeks between the two sessions. In Session 2 participants received albiglutide 50 mg on Day 1 followed by exenatide matching placebo on Day 4. Post-dose MRI was conducted following exenatide matching placebo dose on Day 4 in session 2. Placebo was used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind. Hence, post-exenatide placebo MRI served as the post-albiglutide MRI in this study, to preserve the study blinding and to allow albiglutide sufficient time to reach Tmax.
- Session1 Albiglutide Followed by Session2Off-therapy+Exenatide: Participants received albiglutide 50 mg on Day 1 followed by exenatide matching placebo on Day 4 during Session 1. Post-dose MRI was conducted following exenatide placebo on Day 4 in session 1. There was a wash-out period of 6-9 weeks between the two sessions. In Session 2 participants underwent off-therapy MRI on Day 1 then received albiglutide matching placebo on Day 5 followed by 10 µg of exenatide on Day 8. Post-dose MRI was conducted following exenatide dose on Day 8 in session 2. Placebo was used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind. Hence, post-exenatide placebo MRI served as the post-albiglutide MRI in this study, to preserve the study blinding and to allow albiglutide sufficient time to reach Tmax.
- Session 1 Exenatide Followed by Session2 Off-therapy+Exenatide: Participants received albiglutide matching placebo on Day 1 followed by 10 µg of exenatide on Day 4 during Session 1. Post-dose MRI was conducted following exenatide dose on Day 4 in session 1. There was a wash-out period of 6-9 weeks between the two sessions. In Session 2 participants underwent off-therapy MRI on Day 1 then received albiglutide 50 mg on Day 5 followed by exenatide matching placebo on Day 8. Post-dose MRI was conducted following exenatide matching placebo dose on Day 8 in session 2. Placebo was used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind. Hence, post-exenatide placebo MRI served as the post-albiglutide MRI in this study, to preserve the study blinding and to allow albiglutide sufficient time to reach Tmax.
Period: Session 1 (up to Day 8)
Arm/Group | Session 1 Off-therapy MRI+Albiglutide Followed by Session 2 | Session 1 Off-therapy MRI+Exenatide Followed by Session 2 | Session1 Albiglutide Followed by Session2Off-therapy+Exenatide | Session 1 Exenatide Followed by Session2 Off-therapy+Exenatide
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Wash Out Period (up to Week 9)
Arm/Group | Session 1 Off-therapy MRI+Albiglutide Followed by Session 2 | Session 1 Off-therapy MRI+Exenatide Followed by Session 2 | Session1 Albiglutide Followed by Session2Off-therapy+Exenatide | Session 1 Exenatide Followed by Session2 Off-therapy+Exenatide
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Session 2 (Up to Day 8)
Arm/Group | Session 1 Off-therapy MRI+Albiglutide Followed by Session 2 | Session 1 Off-therapy MRI+Exenatide Followed by Session 2 | Session1 Albiglutide Followed by Session2Off-therapy+Exenatide | Session 1 Exenatide Followed by Session2 Off-therapy+Exenatide
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: Comprised of all participants who received at least one dose of the study treatment.
Groups:
- All Participants: Participants received albiglutide 50 mg or exenatide 10 µg along with matching placebo post off-therapy MRI in a cross-over manner in Session 1 and 2. There was a wash-out period of 6-9 weeks between the two sessions.
Arm/Group | All Participants
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.8 (7.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Mixed Race | 1
  White - Arabic/North African Heritage | 1
  White - White/Caucasian/European Heritage | 2

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygen Level Dependent (BOLD) Signal by Functional Magnetic Resonance Imaging (fMRI) Visual Nauseogenic Task
Description: BOLD signal fMRI Visual Nauseogenic Task data were to be collected at indicated time-points. The seed-to-voxel driven approach included a priori seed Regions of interest (ROIs) placed in brain areas subserving nausea-related processing included regions like interoceptive/sensory (insula, Dorsal anterior cingulate cortex [dACC]), emotional/affective (amygdala, Pregenual anterior cingulate cortex [pgACC]), and cognitive/evaluative (dorsolateral prefrontal cortex [dlPFC]/ Occipitofrontal Circumference [OFC]) brain areas, primary visual (V1) and extrastriate cortices. The primary endpoints of this exploratory study involved combining data from Part A and Part B. The purpose of Part A was decision making for Part B. Placebo was used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind (similar to double dummy), hence data was to be reported in albiglutide, exenatide and off-therapy arms only.
Time Frame: Up to Week 11
Population: All randomized Population (included participants who were randomized to receive study treatment, regardless of whether they took randomized study treatment). Imaging data were analyzed in Part A for only one participant who experienced nausea out of four study participants, and that, as a consequence, data cannot be summarized for Part A.
Groups:
- Albiglutide 50 mg: Participants received albiglutide 50 mg on Day 5 and exenatide placebo on Day 8 or albiglutide 50 mg on Day 1 and exenatide placebo on Day 4 during session 1 or 2 as per randomization. The timing of the albiglutide dose and post-dose MRI were based on the Tmax of albiglutide. Hence, the Day 4 and Day 8 post dose MRI served as the post-albiglutide dose MRI in this study and the exenatide placebo served to preserve the study blinding.
- Exenatide 10 µg: Participants received albiglutide matching placebo on Day 5 and exenatide 10 μg on Day 8 or albiglutide matching placebo on Day 1 and exenatide 10 μg on Day 4 during session 1 or 2 as per randomization schedule. The timing of the exenatide dose and post-dose MRI were based on the Tmax of exentatide. Hence, the Day 4 and Day 8 post dose MRI served as the post exenatide dose MRI and the albiglutide matching placebo served to preserve the study blind.
- Off-therapy MRI: Participants underwent off-therapy MRI. Off-therapy scans served as natural history scan with a 6-9 week washout period between the dosing scans.
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Regional Cerebral Blood Flow (rCBF) by Functional MRI (fMRI)-Arterial Spin Labeling (ASL)
Description: Pseudo-Continuous Arterial spin labeling (pCASL) data were planned to be analyzed to assess rCBF within the brain during using functional MRI scans. Quality control of imaging data were planned to be performed by visual inspection with adequate data denoted by mean rCBF values over the gray matter within a previously defined normal range (i.e., 40-60 millimeter [mm]/100 gram [g] tissue/ minute [min]). In addition, all data were planned to undergo motion and physiological noise correction. Placebo was used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind (similar to double dummy), hence data was reported in albiglutide, exenatide and off-therapy arms only.
Time Frame: Up to Week 11
Population: All randomized Population. Imaging data were analyzed in Part A for only one participant who experienced nausea out of four study participants, and that, as a consequence, data cannot be summarized for Part A.
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Glutamate Concentration in Nausea-associated Brain Regions by Magnetic Resonance Spectroscopy (MRS)
Description: Glutamine/Glutamate (Glx) was planned to be analyzed using proton-density weighted magnetic resonance spectroscopy (1H-MRS). 1H-MRS analysis assessed regional differences in Glx concentrations, normalized as a ratio with creatine. MRS quantification of metabolites of interest were based on frequency domain analysis using a Linear Combination of Model spectra (LCModel). Cramer-Rao lower bounds (CRLBs), as reported from the LCModel analysis, were planned to be used to assess the reliability of the major metabolites and adequate Signal to noise ratio (SNR). CRLBs values less than 40% were further planned to be analyzed. Metabolite maps for each participant, and each session were planned to be calculated. Placebo was used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind (similar to double dummy), hence data was reported in albiglutide, exenatide and off-therapy arms only.
Time Frame: Up to Week 11
Population: as for outcome 2
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Gama-aminobutyric Acid (GABA) Concentration in Nausea-associated Brain Regions by MRS
Description: GABA concentrations was planned to be analyzed using proton-density weighted 1H-MRS. 1H-MRS analysis assessed regional differences GABA concentrations, normalized as a ratio with creatine. MRS quantification of metabolites of interest were based on frequency domain analysis using a LC Model. CRLBs, as reported from the LC Model analysis, were planned to be used to assess the reliability of the major metabolites and adequate SNR. CRLBs values less than 40% were further planned to be analyzed. Metabolite maps for each participant, and each session were planned to be calculated. Placebo was used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind (similar to double dummy), hence data was reported in albiglutide, exenatide and off-therapy arms only.
Time Frame: Up to Week 11
Population: as for outcome 2
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Heart Rate Variability Using Autonomic Response Measures by MRI
Description: Heart rate variability was to be evaluated using autonomic response measure. All peripheral autonomic physiological signals were planned to be collected at 400 Hz using Chart Data Acquisition Software (ADInstruments) on a laptop equipped with a 16-channel Powerlab DAQ System (ADInstruments). Heart rate variability was to be reported as recorded by chart data acquisition software. Placebo was planned to be used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind (similar to double dummy), hence data was reported in albiglutide, exenatide and off-therapy arms only.
Time Frame: Up to Week 11
Population: Safety Population. Imaging data were analyzed in Part A for only one participant who experienced nausea out of four study participants, and that, as a consequence, data cannot be summarized for Part A.
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Intervals Using Autonomic Response Measures by MRI
Description: ECGs intervals were to be evaluated for the participant during the scanning session using autonomic response measures. ECG signal were planned to be collected with an MRI-compatible participant Monitoring system (Biopac 150, Biopac Systems Inc.) through MRI-compatible electrodes (VerMed, Bellows Falls) placed on the chest. Placebo was planned to be used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind (similar to double dummy), hence data was reported in albiglutide, exenatide and off-therapy arms only.
Time Frame: Up to Week 11
Population: as for outcome 5
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormal Respiratory Rate Using Autonomic Response Measures by MRI
Description: Number of participants with abnormal respiratory rate are reported during imaging session was to be evaluated using autonomic response measures. All peripheral autonomic physiological signals were planned to be collected at 400 Hz using Chart Data Acquisition Software (ADInstruments) on a laptop equipped with a 16-channel Powerlab DAQ System (ADInstruments). Placebo was planned to be used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind (similar to double dummy), hence data was reported in albiglutide, exenatide and off-therapy arms only.
Time Frame: Up to Week 11
Population: as for outcome 5
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Skin Conductance Level Using Autonomic Response Measures by MRI
Description: Skin conductance level was to planned to be evaluated with MRI-compatible bipolar Silver (Ag)/Silver chloride (AgCl) finger electrodes placed on the palmar aspect of the second and fourth fingers of the non-dominant (left) hand, prior to the MRI session. All peripheral autonomic physiological signals were planned to be collected at 400 Hz using Chart Data Acquisition Software (ADInstruments) on a laptop equipped with a 16-channel Powerlab DAQ System (ADInstruments). Placebo was planned to be used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind (similar to double dummy), hence data was reported in albiglutide, exenatide and off-therapy arms only.
Time Frame: Up to Week 11
Population: as for outcome 5
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Abnormal Heart Rate for Session 1
Description: Data of participants with abnormal heart rate (measured during site visits by sphygmomanometer) were reported. Participants with low and high heart rate has been presented. Potential clinical concern value for heart rate is < 50 beats per minute to > 120 beats per minute. Safety Population comprised of all participants who received at least one dose of the study treatment.
Time Frame: Day 1: pre-MRI, 0.5 hour post-MRI; Day 4: -2 hours pre-MRI, 0.5 and 1 hour post MRI; Day 5; Day 8: -2 hour pre-MRI, 0.5 and 1 hour post-MRI
Population: Safety Population. Only participants present at specific time points were analyzed. Placebo was planned to be used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, for preserving single-blind (like double dummy), hence data was reported in albiglutide, exenatide and off-therapy arms only
Measure: Count of Participants; unit: Participants
Groups:
- Off-therapy MRI Arm: Participants underwent single off-therapy MRI on Day 1 of session 1 or session 2 as per randomization schedule. Off-therapy scans served as natural history scan with a 6-9 week washout period between the dosing scans. Participants did not undergo MRI on off-therapy visit on Day 5.
- Off-therapy Visit: Participants had out-patient visit on Day 5 for assessment of vital signs. They did not undergo MRI on off-therapy visit on Day 5.
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI Arm | Off-therapy Visit
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants
  Day 1, Pre MRI, high, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  Day 1, Pre MRI, high, n=0, 0, 2, 0 |  |  | 0 |
  Day 1, Pre MRI, low, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  Day 1, Pre MRI, low, n=0, 0, 2, 0 |  |  | 0 |
  Day 1, Post MRI 0.5 hr, high, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  Day 1, Post MRI 0.5 hr, high, n=0, 0, 2, 0 |  |  | 0 |
  Day 1, Post MRI 0.5 hr, low, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  Day 1, Post MRI 0.5 hr, low, n=0, 0, 2, 0 |  |  | 0 |
  Day 4, -2 hr pre-MRI, high, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 4, -2 hr pre-MRI, high, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 4, -2 hr pre-MRI, low, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 4, -2 hr pre-MRI, low, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 4, Post MRI 0.5 hr, high, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 4, Post MRI 0.5 hr, high, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 4, 0.5 hr Post MRI, low, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 4, 0.5 hr Post MRI, low, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 4, 1 hr Post MRI, high, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 4, 1 hr Post MRI, high, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 4, 1 hr Post MRI, low, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 4, 1 hr Post MRI, low, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 5, high, n=0, 0, 0, 2: number analyzed (Participants) | 0 | 0 | 0 | 2
  Day 5, high, n=0, 0, 0, 2 |  |  |  | 0
  Day 5, low, n=0, 0, 0, 2: number analyzed (Participants) | 0 | 0 | 0 | 2
  Day 5, low, n=0, 0, 0, 2 |  |  |  | 0
  Day 8, -2 hr pre-MRI, high, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 8, -2 hr pre-MRI, high, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 8, -2 hr pre-MRI, low, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 8, -2 hr pre-MRI, low, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 8, 0.5 hr Post MRI, high, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 8, 0.5 hr Post MRI, high, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 8, 0.5 hr Post MRI, low, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 8, 0.5 hr Post MRI, low, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 8, 1 hr Post MRI, high, n=0, 1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 8, 1 hr Post MRI, high, n=0, 1, 0, 0 |  | 0 |  |
  Day 8, 1 hr Post MRI, low, n=0, 1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 8, 1 hr Post MRI, low, n=0, 1, 0, 0 |  | 0 |  |

10. Secondary Outcome: Number of Participants With Abnormal Heart Rate for Session 2
Description: Data of participants with abnormal heart rate (measured during site visits by sphygmomanometer) were reported. Participants with low and high heart rate has been presented. Potential clinical concern value for heart rate is < 50 beats per minute to > 120 beats per minute.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI Arm | Off-therapy Visit
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants
  Day 1, Pre MRI, high, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  Day 1, Pre MRI, high, n=0, 0, 2, 0 |  |  | 0 |
  Day 1, Pre MRI, low, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  Day 1, Pre MRI, low, n=0, 0, 2, 0 |  |  | 0 |
  Day 1, Post MRI 0.5 hr, high, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  Day 1, Post MRI 0.5 hr, high, n=0, 0, 2, 0 |  |  | 0 |
  Day 1, Post MRI 0.5 hr, low, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  Day 1, Post MRI 0.5 hr, low, n=0, 0, 2, 0 |  |  | 0 |
  Day 4, -2 hr pre-MRI, high, n=1, 1,0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 4, -2 hr pre-MRI, high, n=1, 1,0, 0 | 0 | 0 |  |
  Day 4, -2 hr pre-MRI, low, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 4, -2 hr pre-MRI, low, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 4, Post MRI 0.5 hr, high, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 4, Post MRI 0.5 hr, high, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 4, 0.5 hr Post MRI, low, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 4, 0.5 hr Post MRI, low, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 4, 1 hr Post MRI, high, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 4, 1 hr Post MRI, high, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 4, 1 hr Post MRI, low, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 4, 1 hr Post MRI, low, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 5, high, n=0, 0, 0, 2: number analyzed (Participants) | 0 | 0 | 0 | 2
  Day 5, high, n=0, 0, 0, 2 |  |  |  | 0
  Day 5, low, n=0, 0, 0, 2: number analyzed (Participants) | 0 | 0 | 0 | 2
  Day 5, low, n=0, 0, 0, 2 |  |  |  | 0
  Day 8, -2 hr pre-MRI, high, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 8, -2 hr pre-MRI, high, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 8, -2 hr pre-MRI, low, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 8, -2 hr pre-MRI, low, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 8, 0.5 hr Post MRI, high, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 8, 0.5 hr Post MRI, high, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 8, 0.5 hr Post MRI, low, n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 8, 0.5 hr Post MRI, low, n=1, 1, 0, 0 | 0 | 0 |  |
  Day 8, 1 hr Post MRI, high, n=0, 1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 8, 1 hr Post MRI, high, n=0, 1, 0, 0 |  | 0 |  |
  Day 8, 1 hr Post MRI, low, n=0, 1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Day 8, 1 hr Post MRI, low, n=0, 1, 0, 0 |  | 0 |  |

11. Secondary Outcome: Number of Participants With Abnormal Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) for Session 1
Description: SBP and DBP were measured in supine position after 5 minutes rest. Data for Session 1 and 2 and for Pre and Post MRI has been presented. Potential clinical concern value for SBP is <100 millimeters of mercury (mmHg) and >170 mmHg. Potential clinical concern value for DBP is <50 mmHg and >110 mmHg.
Time Frame: Day 1: pre-MRI, 0.5 hour post-MRI; Day 4: -2 hours pre-MRI, 0.5 and 1 hour post MRI; Day 5; Day 8: 0.5 and 1 hour post-MRI
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI Arm | Off-therapy Visit
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants
  SBP, Day 1, Pre-MRI, high, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  SBP, Day 1, Pre-MRI, high, n=0, 0, 2, 0 |  |  | 0 |
  SBP, Day 1, Pre-MRI, low, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  SBP, Day 1, Pre-MRI, low, n=0, 0, 2, 0 |  |  | 0 |
  SBP, Day 1, 0.5 hr post MRI, high, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  SBP, Day 1, 0.5 hr post MRI, high, n=0, 0, 2, 0 |  |  | 0 |
  SBP, Day 1,0.5 hr post MRI , low, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  SBP, Day 1,0.5 hr post MRI , low, n=0, 0, 2, 0 |  |  | 0 |
  SBP, Day 4,-2 hr pre-MRI, high, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 4,-2 hr pre-MRI, high, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 4,-2 hr pre-MRI, low, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 4,-2 hr pre-MRI, low, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 4,0.5 hr post MRI , high, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 4,0.5 hr post MRI , high, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 4,0.5 hr post MRI, low, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 4,0.5 hr post MRI, low, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 4,1 hr post MRI , high, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 4,1 hr post MRI , high, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 4,1 hr post MRI , low, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 4,1 hr post MRI , low, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 5, high, n=0, 0, 0, 2: number analyzed (Participants) | 0 | 0 | 0 | 2
  SBP, Day 5, high, n=0, 0, 0, 2 |  |  |  | 0
  SBP, Day 5, low, n=0, 0, 0, 2: number analyzed (Participants) | 0 | 0 | 0 | 2
  SBP, Day 5, low, n=0, 0, 0, 2 |  |  |  | 0
  SBP, Day 8,0.5 hr Post MRI, high, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 8,0.5 hr Post MRI, high, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 8,0.5 hr Post MRI, low, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 8,0.5 hr Post MRI, low, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 8,1 hr Post MRI, high, n= 0,1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  SBP, Day 8,1 hr Post MRI, high, n= 0,1, 0, 0 |  | 0 |  |
  SBP, Day 8,1 hr post MRI , low, n= 0,1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  SBP, Day 8,1 hr post MRI , low, n= 0,1, 0, 0 |  | 0 |  |
  DBP, Day 1, Pre MRI, high,n= 0,0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  DBP, Day 1, Pre MRI, high,n= 0,0, 2, 0 |  |  | 0 |
  DBP, Day 1, Pre MRI, low,n= 0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  DBP, Day 1, Pre MRI, low,n= 0, 0, 2, 0 |  |  | 0 |
  DBP, Day 1,0.5 hr post MRI, high,n= 0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  DBP, Day 1,0.5 hr post MRI, high,n= 0, 0, 2, 0 |  |  | 0 |
  DBP, Day 1,0.5 hr post MRI, low,n= 0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  DBP, Day 1,0.5 hr post MRI, low,n= 0, 0, 2, 0 |  |  | 0 |
  DBP, Day 4,-2 hr pre-MRI, high, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 4,-2 hr pre-MRI, high, n=1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 4,-2 hr pre-MRI, low, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 4,-2 hr pre-MRI, low, n=1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 4,0.5 hr Post MRI, high,n= 1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 4,0.5 hr Post MRI, high,n= 1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 4,0.5 hr Post MRI, low,n= 1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 4,0.5 hr Post MRI, low,n= 1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 4,1 hr post MRI, high,n= 1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 4,1 hr post MRI, high,n= 1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 4,1 hr post MRI , low,n= 1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 4,1 hr post MRI , low,n= 1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 5, high, n= 0,0,0,2: number analyzed (Participants) | 0 | 0 | 0 | 2
  DBP, Day 5, high, n= 0,0,0,2 |  |  |  | 0
  DBP, Day 5, low, n= 0,0,0,2: number analyzed (Participants) | 0 | 0 | 0 | 2
  DBP, Day 5, low, n= 0,0,0,2 |  |  |  | 0
  DBP, Day 8, 0.5 hr post MRI ,high, n=1,1,0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 8, 0.5 hr post MRI ,high, n=1,1,0, 0 | 0 | 0 |  |
  DBP, Day 8, 0.5 hr post MRI, low, n= 1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 8, 0.5 hr post MRI, low, n= 1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 8, 1 hr post MRI, high, n=0,1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  DBP, Day 8, 1 hr post MRI, high, n=0,1, 0, 0 |  | 0 |  |
  DBP, Day 8, 1 hr post MRI, low, n=0,1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  DBP, Day 8, 1 hr post MRI, low, n=0,1, 0, 0 |  | 0 |  |

12. Secondary Outcome: Number of Participants With Abnormal SBP and DBP for Session 2
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI | Off-therapy Visit
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants
  SBP, Day 1, Pre-MRI, high, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  SBP, Day 1, Pre-MRI, high, n=0, 0, 2, 0 |  |  | 0 |
  SBP, Day 1, Pre-MRI, low, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  SBP, Day 1, Pre-MRI, low, n=0, 0, 2, 0 |  |  | 0 |
  SBP, Day 1, 0.5 hr post MRI, high, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  SBP, Day 1, 0.5 hr post MRI, high, n=0, 0, 2, 0 |  |  | 0 |
  SBP, Day 1,0.5 hr post MRI , low, n=0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  SBP, Day 1,0.5 hr post MRI , low, n=0, 0, 2, 0 |  |  | 0 |
  SBP, Day 4,-2 hr pre-MRI, high, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 4,-2 hr pre-MRI, high, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 4,-2 hr pre-MRI, low, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 4,-2 hr pre-MRI, low, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 4,0.5 hr post MRI , high, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 4,0.5 hr post MRI , high, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 4,0.5 hr post MRI, low, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 4,0.5 hr post MRI, low, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 4,1 hr post MRI , high, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 4,1 hr post MRI , high, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 4,1 hr post MRI , low, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 4,1 hr post MRI , low, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 5, high, n=0, 0, 0, 2: number analyzed (Participants) | 0 | 0 | 0 | 2
  SBP, Day 5, high, n=0, 0, 0, 2 |  |  |  | 0
  SBP, Day 5, low, n=0, 0, 0, 2: number analyzed (Participants) | 0 | 0 | 0 | 2
  SBP, Day 5, low, n=0, 0, 0, 2 |  |  |  | 0
  SBP, Day 8,0.5 hr Post MRI, high, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 8,0.5 hr Post MRI, high, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 8,0.5 hr Post MRI, low, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  SBP, Day 8,0.5 hr Post MRI, low, n=1,1, 0, 0 | 0 | 0 |  |
  SBP, Day 8,1 hr Post MRI, high, n= 0,1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  SBP, Day 8,1 hr Post MRI, high, n= 0,1, 0, 0 |  | 0 |  |
  SBP, Day 8,1 hr post MRI , low, n= 0,1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  SBP, Day 8,1 hr post MRI , low, n= 0,1, 0, 0 |  | 0 |  |
  DBP, Day 1, Pre MRI, high,n= 0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  DBP, Day 1, Pre MRI, high,n= 0, 0, 2, 0 |  |  | 0 |
  DBP, Day 1, Pre MRI, low,n= 0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  DBP, Day 1, Pre MRI, low,n= 0, 0, 2, 0 |  |  | 0 |
  DBP, Day 1,0.5 hr post MRI, high,n= 0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  DBP, Day 1,0.5 hr post MRI, high,n= 0, 0, 2, 0 |  |  | 1 |
  DBP, Day 1,0.5 hr post MRI, low,n= 0, 0, 2, 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  DBP, Day 1,0.5 hr post MRI, low,n= 0, 0, 2, 0 |  |  | 0 |
  DBP, Day 4,-2 hr pre-MRI, high, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 4,-2 hr pre-MRI, high, n=1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 4,-2 hr pre-MRI, low, n=1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 4,-2 hr pre-MRI, low, n=1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 4,0.5 hr Post MRI, high,n= 1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 4,0.5 hr Post MRI, high,n= 1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 4,0.5 hr Post MRI, low,n= 1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 4,0.5 hr Post MRI, low,n= 1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 4,1 hr post MRI, high,n= 1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 4,1 hr post MRI, high,n= 1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 4,1 hr post MRI , low,n= 1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 4,1 hr post MRI , low,n= 1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 5, high, n= 0,0,0,2: number analyzed (Participants) | 0 | 0 | 0 | 2
  DBP, Day 5, high, n= 0,0,0,2 |  |  |  | 0
  DBP, Day 5, low, n= 0,0,0,2: number analyzed (Participants) | 0 | 0 | 0 | 2
  DBP, Day 5, low, n= 0,0,0,2 |  |  |  | 0
  DBP, Day 8, 0.5 hr post MRI ,high, n=1,1,0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 8, 0.5 hr post MRI ,high, n=1,1,0, 0 | 0 | 0 |  |
  DBP, Day 8, 0.5 hr post MRI, low, n= 1,1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  DBP, Day 8, 0.5 hr post MRI, low, n= 1,1, 0, 0 | 0 | 0 |  |
  DBP, Day 8, 1 hr post MRI, high, n=0,1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  DBP, Day 8, 1 hr post MRI, high, n=0,1, 0, 0 |  | 0 |  |
  DBP, Day 8, 1 hr post MRI, low, n=0,1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  DBP, Day 8, 1 hr post MRI, low, n=0,1, 0, 0 |  | 0 |  |

13. Secondary Outcome: Number of Participants With Abnormal Clinical Chemistry Parameters
Description: Clinical chemistry parameters included assessment of blood urea nitrogen (BUN), creatinine, epidermal growth factor receptor (eGRF), potassium, sodium, calcium, Aspartate transaminase (AST), Alanine transaminase (AST), Alkaline phosphatase, total and direct bilirubin, total protein and albumin.
Time Frame: Up to Week 11
Population: Safety Population. The data was reported in cumulative format as placebo was included to maintain the single blind only; similar to double dummy.
Measure: Count of Participants; unit: Participants
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Abnormal Hematology Parameters
Description: Hematology parameters included assessment of platelet count, red blood cell (RBC) count, hemoglobin, hemotocrit, RBC indices including mean corpuscular volume and mean corpuscular hemoglobin (MCH), and White blood cells (WBC) count with differential count including, neutrophils, lymphocytes, monocytes, eosinophils and basophils.
Time Frame: Up to Week 11
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

15. Secondary Outcome: Number of Participants With Abnormal Urinalysis
Description: Urinalysis parameters included assessment of specific gravity, microscopic analysis, and potential of hydrogen (pH), glucose, protein, blood and ketones by dipstick method.
Time Frame: Up to Week 11
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With Abnormal Glycemic Parameters
Description: Glycemic parameters included assessment of capillary blood glucose and fasting plasma glucose.
Time Frame: Up to Week 11
Population: Safety Population.The data was reported in cumulative format as placebo was included to maintain the single blind only; similar to double dummy.
Measure: Count of Participants; unit: Participants
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

17. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AE) With Incidence > = 2 % and Serious AEs (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment were categorized as SAE. Data of participants with non-serious AEs ( with incidence >= 2%) and SAEs has been presented. Placebo was included to maintain the single blind only; similar to double dummy.
Time Frame: Up to Week 13
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Albiglutide Matching Placebo: Participants in Session 1 received albiglutide matching placebo on Day 1 or Day 5 and during Session 2 participants received albiglutide matching placebo on Day 5 or Day 1. Placebo was used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind. Hence, post-exenatide placebo MRI served as the post-albiglutide MRI in this study, to preserve the study blinding and to allow albiglutide sufficient time to reach Tmax.
- Exenatide Matching Placebo: Participants in Session 1 received exenatide matching placebo on Day 4 or Day 8 and during Session 2 participants received exenatide matching placebo on Day 8 or Day 4. Placebo was used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind. Hence, post-exenatide placebo MRI served as the post-albiglutide MRI in this study, to preserve the study blinding and to allow albiglutide sufficient time to reach Tmax.
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Albiglutide Matching Placebo | Exenatide Matching Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4
Participants
  Non-serious AEs | 1 | 0 | 0 | 0
  SAE | 0 | 0 | 0 | 0

18. Secondary Outcome: Nausea Ratings Scale to Rate Nausea Sensation Using Autonomic Response Measures by MRI
Description: Nausea ratings were planned to be collected during motion sickness provocation using a 0-4 numerical rating scale (NRS), where 1 is rated as minimal nausea experienced and 4 as severe nausea was experienced. Participants were asked to press buttons on a MRI compatible button-box to rate nausea from 0 to 4. Placebo was planned to be used to enable albiglutide and exenatide to be dosed at different times relative to MRI due to differences in Tmax, while preserving single-blind (similar to double dummy), hence data was reported in albiglutide, exenatide and off-therapy arms only.
Time Frame: Up to Week 11
Population: as for outcome 5
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Gastrointestinal (GI) Visual Analogue Scale (VAS) for Assessment of Nausea for Session 1
Description: Participant completed VAS to record their perception of stomach fullness, hunger, nausea, bloating and abdominal pain. The VAS was represented by lines, 100 millimeter in length, anchored with words describing the most negative rating on the left and the most positive rating on the right. Scores ranged from 0 mm to 100 mm. Scores of 0 mm are worst (most negative rating on the left) and scores of 100 mm are best (most positive rating on the right). NA indicates that data were not available as standard deviation could not be calculated due to low number of participants.
Time Frame: Day 1 (Pre-MRI and 0.5 hour post-MRI); Day 4 (Pre-MRI and 0.5 hour post-MRI); and Day 8 (Pre-MRI and 0.5 hour post-MRI)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 2 | 2 | 2
Scores on scale
  Hunger, Day1, pre-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Hunger, Day1, pre-MRI,n=0,0,2 |  |  | 29.0 (41.01)
  Hunger, Day1, 0.5 hour post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Hunger, Day1, 0.5 hour post-MRI,n=0,0,2 |  |  | 55.0 (21.21)
  Hunger, Day4, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Hunger, Day4, pre-MRI,n=1,1,0 | 65.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 40.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Hunger, Day4, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Hunger, Day4, 0.5 hour post-MRI,n=1,1,0 | 66.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 50.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Hunger, Day8, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Hunger, Day8, pre-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 25.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Hunger, Day8, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Hunger, Day8, 0.5 hour post-MRI,n=1,1,0 | 31.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 26.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Stomach fullness, Day1, pre-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Stomach fullness, Day1, pre-MRI,n=0,0,2 |  |  | 9.0 (9.90)
  Stomach fullness, Day1, 0.5 hour post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Stomach fullness, Day1, 0.5 hour post-MRI,n=0,0,2 |  |  | 0.5 (0.71)
  Stomach fullness, Day4,pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Stomach fullness, Day4,pre-MRI,n=1,1,0 | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Stomach fullness, Day4, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Stomach fullness, Day4, 0.5 hour post-MRI,n=1,1,0 | 6.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Stomach fullness, Day8, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Stomach fullness, Day8, pre-MRI,n=1,1,0 | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Stomach fullness, Day8, 0.5 hour post- MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Stomach fullness, Day8, 0.5 hour post- MRI,n=1,1,0 | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Nausea, Day1, pre- MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Nausea, Day1, pre- MRI,n=0,0,2 |  |  | 1.0 (1.41)
  Nausea, Day1,0.5 hour post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Nausea, Day1,0.5 hour post-MRI,n=0,0,2 |  |  | 19.0 (25.46)
  Nausea, Day4, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Nausea, Day4, pre-MRI,n=1,1,0 | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Nausea, Day4, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Nausea, Day4, 0.5 hour post-MRI,n=1,1,0 | 24.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Nausea, Day8, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Nausea, Day8, pre-MRI,n=1,1,0 | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Nausea, Day8,0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Nausea, Day8,0.5 hour post-MRI,n=1,1,0 | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Bloating, Day1, pre-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Bloating, Day1, pre-MRI,n=0,0,2 |  |  | 1.5 (0.71)
  Bloating, Day1, 0.5 hour post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Bloating, Day1, 0.5 hour post-MRI,n=0,0,2 |  |  | 1.0 (1.41)
  Bloating, Day4, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Bloating, Day4, pre-MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Bloating, Day4, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Bloating, Day4, 0.5 hour post-MRI,n=1,1,0 | 4.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Bloating, Day8, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Bloating, Day8, pre-MRI,n=1,1,0 | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Bloating, Day8, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Bloating, Day8, 0.5 hour post-MRI,n=1,1,0 | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Abdominal pain, Day1, pre-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Abdominal pain, Day1, pre-MRI,n=0,0,2 |  |  | 2.0 (1.41)
  Abdominal pain, Day1,0.5 hour post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Abdominal pain, Day1,0.5 hour post-MRI,n=0,0,2 |  |  | 1.5 (2.12)
  Abdominal pain, Day4, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Abdominal pain, Day4, pre-MRI,n=1,1,0 | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Abdominal pain, Day4, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Abdominal pain, Day4, 0.5 hour post-MRI,n=1,1,0 | 5.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Abdominal pain, Day8, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Abdominal pain, Day8, pre-MRI,n=1,1,0 | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Abdominal pain, Day8, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Abdominal pain, Day8, 0.5 hour post-MRI,n=1,1,0 | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |

20. Secondary Outcome: GI VAS for Assessment of Nausea for Session 2
Description: as for outcome 19
Time Frame: Day 1 (Pre-MRI and 0.5 hour post-MRI); Day 4 (Pre-MRI and 0.5 hour post-MRI); and Day 8 (Pre-MRI and 0.5 hour post-MRI)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 2 | 2 | 2
Scores on scale
  Hunger, Day1, pre-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Hunger, Day1, pre-MRI,n=0,0,2 |  |  | 54.5 (33.23)
  Hunger, Day1,0.5 hour post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Hunger, Day1,0.5 hour post-MRI,n=0,0,2 |  |  | 67.5 (23.33)
  Hunger, Day4, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Hunger, Day4, pre-MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 53.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Hunger, Day4,0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Hunger, Day4,0.5 hour post-MRI,n=1,1,0 | 57.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 66.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Hunger, Day8, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Hunger, Day8, pre-MRI,n=1,1,0 | 38.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 77.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Hunger, Day8, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Hunger, Day8, 0.5 hour post-MRI,n=1,1,0 | 53.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 73.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Stomach fullness, Day1, pre-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Stomach fullness, Day1, pre-MRI,n=0,0,2 |  |  | 11.5 (4.95)
  Stomach fullness, Day1, 0.5 hour post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Stomach fullness, Day1, 0.5 hour post-MRI,n=0,0,2 |  |  | 7.0 (7.07)
  Stomach fullness, Day4, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Stomach fullness, Day4, pre-MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Stomach fullness, Day4,0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Stomach fullness, Day4,0.5 hour post-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Stomach fullness, Day8, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Stomach fullness, Day8, pre-MRI,n=1,1,0 | 11.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 10.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Stomach fullness, Day8,0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Stomach fullness, Day8,0.5 hour post-MRI,n=1,1,0 | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 13.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Nausea, Day1, pre-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Nausea, Day1, pre-MRI,n=0,0,2 |  |  | 23.5 (31.82)
  Nausea, Day1, 0.5 hour post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Nausea, Day1, 0.5 hour post-MRI,n=0,0,2 |  |  | 17.5 (14.85)
  Nausea, Day4, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Nausea, Day4, pre-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Nausea, Day4,0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Nausea, Day4,0.5 hour post-MRI,n=1,1,0 | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Nausea, Day8, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Nausea, Day8, pre-MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 48.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Nausea, Day8, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Nausea, Day8, 0.5 hour post-MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 38.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Bloating, Day1, pre-MRI,n=0, 0, 2: number analyzed (Participants) | 0 | 0 | 2
  Bloating, Day1, pre-MRI,n=0, 0, 2 |  |  | 6.0 (7.07)
  Bloating, Day1, 0.5 hour post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Bloating, Day1, 0.5 hour post-MRI,n=0,0,2 |  |  | 4.0 (4.24)
  Bloating, Day4, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Bloating, Day4, pre-MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Bloating, Day4,0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Bloating, Day4,0.5 hour post-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Bloating, Day8, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Bloating, Day8, pre-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 6.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Bloating, Day8, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Bloating, Day8, 0.5 hour post-MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 6.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Abdominal pain, Day1, pre-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Abdominal pain, Day1, pre-MRI,n=0,0,2 |  |  | 7.5 (9.19)
  Abdominal pain, Day1, 0.5 hour post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  Abdominal pain, Day1, 0.5 hour post-MRI,n=0,0,2 |  |  | 4.0 (4.24)
  Abdominal pain, Day4, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Abdominal pain, Day4, pre-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Abdominal pain, Day4, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Abdominal pain, Day4, 0.5 hour post-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 0.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Abdominal pain, Day8, pre-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Abdominal pain, Day8, pre-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 7.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  Abdominal pain, Day8, 0.5 hour post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  Abdominal pain, Day8, 0.5 hour post-MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 6.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |

21. Secondary Outcome: Motion Sickness Assessment Questionnaire (MSAQ) for Assessment of Nausea for Session 1
Description: Participant completed MSAQ to quantify the severity of different dimensions of nausea induced by motion sickness. There were total 16 items: 4 related to gastro-intestinal (GI), 5 related to central (C), 3 related to peripheral (P) and 4 related to sopite-related (SR). All items were scored individually on a scale of 1-9 where 1 means 'not at all severe' and 9 means 'severe', with higher score indicates more severity. Individual 16 items with their scores are presented. NA indicates that data were not available as standard deviation could not be calculated due to low number of participants.
Time Frame: Day 1 0.5 hour post-MRI; Day 4 0.5 hour post-MRI; and Day 8 0.5 hour post-MRI
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 2 | 2 | 2
Scores on scale
  C, Felt faint like, Day1,0.5 hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  C, Felt faint like, Day1,0.5 hr,Post MRI,n=0,0,2 |  |  | 4.0 (4.24)
  C, Felt faint like, Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt faint like, Day4,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt faint like, Day8, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt faint like, Day8, 0.5 hr,Post MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt lightheaded, Day1,0.5 hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  C, Felt lightheaded, Day1,0.5 hr,Post MRI,n=0,0,2 |  |  | 5.5 (3.54)
  C, Felt lightheaded, Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt lightheaded, Day4,0.5 hr,Post MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt lightheaded, Day8, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt lightheaded, Day8, 0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt disoriented, Day1,0.5 hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  C, Felt disoriented, Day1,0.5 hr,Post MRI,n=0,0,2 |  |  | 4.5 (2.12)
  C, Felt disoriented, Day4, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt disoriented, Day4, 0.5 hr,Post MRI,n=1,1,0 | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt disoriented, Day8, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt disoriented, Day8, 0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt dizzy, Day1,0.5 hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  C, Felt dizzy, Day1,0.5 hr,Post MRI,n=0,0,2 |  |  | 8.0 (1.41)
  C, Felt dizzy, Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt dizzy, Day4,0.5 hr,Post MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt dizzy, Day8,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt dizzy, Day8,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt spinning, Day1,0.5 hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  C, Felt spinning, Day1,0.5 hr,Post MRI,n=0,0,2 |  |  | 5.5 (4.95)
  C, Felt spinning, Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt spinning, Day4,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt spinning, Day8, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt spinning, Day8, 0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, stomach sick, Day1,0.5hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  GI, stomach sick, Day1,0.5hr,Post MRI,n=0,0,2 |  |  | 5.0 (4.24)
  GI, stomach sick, Day4,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, stomach sick, Day4,0.5hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, stomach sick, Day8,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, stomach sick, Day8,0.5hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, felt queasy, Day1,0.5hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  GI, felt queasy, Day1,0.5hr,Post MRI,n=0,0,2 |  |  | 6.5 (2.12)
  GI, felt queasy, Day4,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, felt queasy, Day4,0.5hr,Post MRI,n=1,1,0 | 4.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, felt queasy, Day8,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, felt queasy, Day8,0.5hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, nauseated, Day1, 0.5hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  GI, nauseated, Day1, 0.5hr,Post MRI,n=0,0,2 |  |  | 6.5 (2.12)
  GI, nauseated, Day4,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, nauseated, Day4,0.5hr,Post MRI,n=1,1,0 | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, nauseated, Day8,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, nauseated, Day8,0.5hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, may vomit, Day1,0.5hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  GI, may vomit, Day1,0.5hr,Post MRI,n=0,0,2 |  |  | 6.5 (2.12)
  GI, may vomit, Day4,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, may vomit, Day4,0.5hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, may vomit, Day8,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, may vomit, Day8,0.5hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  P, sweaty, Day1,0.5hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  P, sweaty, Day1,0.5hr,Post MRI,n=0,0,2 |  |  | 4.5 (4.95)
  P, sweaty, Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  P, sweaty, Day4,0.5 hr,Post MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  P, sweaty, Day8, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  P, sweaty, Day8, 0.5 hr,Post MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  P, clammy/cold sweat,Day1,0.5hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  P, clammy/cold sweat,Day1,0.5hr,Post MRI,n=0,0,2 |  |  | 4.5 (4.95)
  P,clammy/cold sweat,Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  P,clammy/cold sweat,Day4,0.5 hr,Post MRI,n=1,1,0 | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  P, clammy/cold sweat,Day8,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  P, clammy/cold sweat,Day8,0.5 hr,Post MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  P, hot/warm, Day1,0.5hr,Post MRI,n=0, 0, 2: number analyzed (Participants) | 0 | 0 | 2
  P, hot/warm, Day1,0.5hr,Post MRI,n=0, 0, 2 |  |  | 2.5 (2.12)
  P, hot/warm, Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  P, hot/warm, Day4,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  P, hot/warm, Day8, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  P, hot/warm, Day8, 0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR,annoyed/irritated,Day1,0.5hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  SR,annoyed/irritated,Day1,0.5hr,Post MRI,n=0,0,2 |  |  | 5.0 (4.24)
  SR,annoyed/irritated,Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR,annoyed/irritated,Day4,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR,annoyed/irritated,Day8, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR,annoyed/irritated,Day8, 0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR, drowsy, Day1,0.5hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  SR, drowsy, Day1,0.5hr,Post MRI,n=0,0,2 |  |  | 1.0 (0.00)
  SR, drowsy, Day4, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR, drowsy, Day4, 0.5 hr,Post MRI,n=1,1,0 | 5.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR, drowsy, Day8, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR, drowsy, Day8, 0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR, tired/fatigued, Day1,0.5hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  SR, tired/fatigued, Day1,0.5hr,Post MRI,n=0,0,2 |  |  | 1.5 (0.71)
  SR, tired/fatigued, Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR, tired/fatigued, Day4,0.5 hr,Post MRI,n=1,1,0 | 4.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR, tired/fatigued, Day8,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR, tired/fatigued, Day8,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR, uneasy, Day1,0.5hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  SR, uneasy, Day1,0.5hr,Post MRI,n=0,0,2 |  |  | 8.0 (0.00)
  SR, uneasy, Day4, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR, uneasy, Day4, 0.5 hr,Post MRI,n=1,1,0 | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR, uneasy, Day8,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR, uneasy, Day8,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |

22. Secondary Outcome: MSAQ for Assessment of Nausea for Session 2
Description: as for outcome 21
Time Frame: Day 1 0.5 hour post-MRI; Day 4 0.5 hour post-MRI; and Day 8 0.5 hour post-MRI
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Off-therapy MRI
Number analyzed (Participants) | 2 | 2 | 2
Scores on scale
  C, Felt faint like, Day1,0.5 hr Post MRI ,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  C, Felt faint like, Day1,0.5 hr Post MRI ,n=0,0,2 |  |  | 3.0 (2.83)
  C, Felt faint like, Day4,0.5 hr Post MRI ,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt faint like, Day4,0.5 hr Post MRI ,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt faint like, Day8,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt faint like, Day8,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt lightheaded, Day1,0.5 hr Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  C, Felt lightheaded, Day1,0.5 hr Post MRI,n=0,0,2 |  |  | 2.0 (0.00)
  C, Felt lightheaded, Day4, 0.5 hr Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt lightheaded, Day4, 0.5 hr Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt lightheaded, Day8, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt lightheaded, Day8, 0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt disoriented, Day1,0.5 hr, Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  C, Felt disoriented, Day1,0.5 hr, Post MRI,n=0,0,2 |  |  | 2.0 (1.41)
  C, Felt disoriented, Day4,0.5 hr Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt disoriented, Day4,0.5 hr Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt disoriented, Day8,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt disoriented, Day8,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt dizzy, Day1, 0.5 hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  C, Felt dizzy, Day1, 0.5 hr,Post MRI,n=0,0,2 |  |  | 2.0 (0.00)
  C, Felt dizzy, Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt dizzy, Day4,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt dizzy, Day8,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt dizzy, Day8,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt spinning, Day1,0.5 hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  C, Felt spinning, Day1,0.5 hr,Post MRI,n=0,0,2 |  |  | 4.0 (4.24)
  C, Felt spinning, Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt spinning, Day4,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  C, Felt spinning, Day8,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  C, Felt spinning, Day8,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, stomach sick, Day1,0.5hr,Post MRI, n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  GI, stomach sick, Day1,0.5hr,Post MRI, n=0,0,2 |  |  | 5.0 (0.00)
  GI, stomach sick, Day4, 0.5hr post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, stomach sick, Day4, 0.5hr post-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, stomach sick, Day8,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, stomach sick, Day8,0.5hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, felt queasy, Day1, 0.5hr post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  GI, felt queasy, Day1, 0.5hr post-MRI,n=0,0,2 |  |  | 4.5 (2.12)
  GI, felt queasy, Day4,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, felt queasy, Day4,0.5hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, felt queasy, Day8, 0.5h,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, felt queasy, Day8, 0.5h,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 2.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, nauseated, Day1,0.5hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  GI, nauseated, Day1,0.5hr,Post MRI,n=0,0,2 |  |  | 6.0 (1.41)
  GI, nauseated, Day4,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, nauseated, Day4,0.5hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, nauseated, Day8,0.5hr,Post MRI, n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, nauseated, Day8,0.5hr,Post MRI, n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, may vomit, Day1,0.5hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  GI, may vomit, Day1,0.5hr,Post MRI,n=0,0,2 |  |  | 2.0 (0.00)
  GI, may vomit, Day4,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, may vomit, Day4,0.5hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  GI, may vomit, Day8,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  GI, may vomit, Day8,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  P, sweaty, Day1,0.5 hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  P, sweaty, Day1,0.5 hr,Post MRI,n=0,0,2 |  |  | 1.5 (0.71)
  P, sweaty, Day4, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  P, sweaty, Day4, 0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  P, sweaty, Day8,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  P, sweaty, Day8,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  P,clammy/cold sweat,Day1,0.5hr,post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  P,clammy/cold sweat,Day1,0.5hr,post-MRI,n=0,0,2 |  |  | 2.0 (1.41)
  P, clammy/cold sweat, Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  P, clammy/cold sweat, Day4,0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  P,clammy/cold sweat,Day8,0.5hr,Post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  P,clammy/cold sweat,Day8,0.5hr,Post-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  P, hot/warm, Day1,0.5 hr, Post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  P, hot/warm, Day1,0.5 hr, Post-MRI,n=0,0,2 |  |  | 1.0 (0.00)
  P, hot/warm, Day4, 0.5 hr,Post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  P, hot/warm, Day4, 0.5 hr,Post-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  P, hot/warm,Day8, 0.5 hr Post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  P, hot/warm,Day8, 0.5 hr Post-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR,annoyed/irritated,Day1,0.5hr, Post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  SR,annoyed/irritated,Day1,0.5hr, Post-MRI,n=0,0,2 |  |  | 1.5 (0.71)
  SR,annoyed/irritated,Day4,0.5hr,Post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR,annoyed/irritated,Day4,0.5hr,Post-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR,annoyed/irritated,Day8,0.5hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR,annoyed/irritated,Day8,0.5hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR, drowsy, Day1, 0.5 hr,Post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  SR, drowsy, Day1, 0.5 hr,Post-MRI,n=0,0,2 |  |  | 4.0 (1.41)
  SR, drowsy, Day4, 0.5 hr,Post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR, drowsy, Day4, 0.5 hr,Post-MRI,n=1,1,0 | 5.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR, drowsy, Day8, 0.5 hr, Post-MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR, drowsy, Day8, 0.5 hr, Post-MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 5.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR, tired/fatigued, Day1,0.5 hr,Post MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  SR, tired/fatigued, Day1,0.5 hr,Post MRI,n=0,0,2 |  |  | 4.5 (3.54)
  SR, tired/fatigued, Day4,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR, tired/fatigued, Day4,0.5 hr,Post MRI,n=1,1,0 | 4.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR, tired/fatigued, Day8,0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR, tired/fatigued, Day8,0.5 hr,Post MRI,n=1,1,0 | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 3.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR, uneasy, Day1, 0.5 hr,Post-MRI,n=0,0,2: number analyzed (Participants) | 0 | 0 | 2
  SR, uneasy, Day1, 0.5 hr,Post-MRI,n=0,0,2 |  |  | 4.0 (2.83)
  SR, uneasy, Day4, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR, uneasy, Day4, 0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |
  SR, uneasy, Day8, 0.5 hr,Post MRI,n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  SR, uneasy, Day8, 0.5 hr,Post MRI,n=1,1,0 | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. | 1.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated due to low number of participants. |

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study treatment up to Week 13.
Description: SAEs and Non-serious AEs for participants of Safety Population were reported. AEs data was reported per Intervention.
Groups:
- Albiglutide Matching Placebo: Participants in Session 1 received albiglutide matching placebo on Day 1 and during Session 2 participants received albiglutide matching placebo on Day 5. There was a wash-out period of 6-9 weeks between the two sessions.
- Exenatide Matching Placebo: Participants in Session 1 received exenatide matching placebo on Day 4 and during Session 2 participants received exenatide matching placebo on Day 8. There was a wash-out period of 6-9 weeks between the two sessions.
Arm/Group | Albiglutide 50 mg | Exenatide 10 µg | Albiglutide Matching Placebo | Exenatide Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 0/4 | 0/4 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albiglutide 50 mg (N=4) | Exenatide 10 µg (N=4) | Albiglutide Matching Placebo (N=4) | Exenatide Matching Placebo (N=4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT02802514/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT02802514/SAP_001.pdf